CLINICAL TRIAL: NCT07065513
Title: Effects of High Energy Nutritional Protein Based Bar on Performance of Young Athletes
Brief Title: Effects of High-energy Nutritional Protein-based Bar on the Performance of Young Athletes
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: MSAHSW/Batch-Fall23/927
Record Dates: First submitted 2025-06-28; First posted 2025-07-15 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Enduring Personality Change

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Normal diet (Experimental)
  Interventions: Diagnostic Test: Normal diet
- Normal diet plus nutritional protein-based bar (Experimental)
  Interventions: Combination Product: Normal diet plus nutritional protein-based bar

INTERVENTIONS:
Diagnostic Test: Normal diet — Normal diet (control group, 20 participants: 10 boys and 10 girls).
  Arms: Normal diet
Combination Product: Normal diet plus nutritional protein-based bar — : Normal diet plus nutritional protein-based bar (intervention group, 20 participants: 10 boys and 10 girls). The participants will consume 3 servings of 14g each per day, providing 6.8g protein and 283 kcal
  Arms: Normal diet plus nutritional protein-based bar

SUMMARY:
A study will be conducted in Lahore. Non probability convenience sampling technique will be applied on patients who will be allocated through computerized randomization into group A & group B to collect data.

DETAILED DESCRIPTION:
Group A will be given normal diet and group B will be given normal diet in addition to protein bars. The study will be completed within the time duration of nine months. Primary Outcome measures of the research will be protein effects and quality of life in protein deficiency malnourished children. Data will be analyzed using SPSS software version 25.

ELIGIBILITY:
Inclusion Criteria:

* Boys and girls aged 18-25 years.
* Regularly playing team sports (football, volleyball, cricket).
* Average of 5 hours per day spent in field activities (practice + matches).

Exclusion Criteria:

* Allergies to bar ingredients (e.g., nuts).
* Metabolic disorders affecting nutrient absorption.
* Protein-energy malnutrition (PEM).
* Hospitalized adults.
* Eating disorders or diagnosed mental illness"

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Self-Administered Questionnaire | 12 Months
  Self-Administered Questionnaire for getting different values and measurements according to the healthcare values to check the nutritional effects on the body

CONTACTS AND LOCATIONS:
Locations (1):
- Lahore sports complex, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No